CLINICAL TRIAL: NCT04687345
Title: Clinical Research of Using Lateral Supramalleolar Perforator Flap Reconstruction Through Branches Outside of the Ankle Tissue Defects
Brief Title: Lateral Supramalleolar Perforator Flap Reconstruction Through Branches Outside of the Ankle Tissue Defects
Status: Completed | Type: Observational
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Shih Yu-Jen, Lecturer/Attending Doctor, National Defense Medical Center, Taiwan
Other Study IDs: PerforatorFlap2018
Record Dates: First submitted 2020-12-08; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Ankle Tissue Injury Wound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Propeller Flap: The propeller flap is based on a perforator that serves as a pivot joint, allowing the flap to rotate up to 180°. It provides the advantages of greater freedom of movement and versatility in flap design.
- Rotation Flap: The rotation flap is primarily supplied by the perforator artery accompanied by the random supply from the skin base. It is also associated with a lower venous congestion risk.

SUMMARY:
The lateral ankle is a common site of tissue defects and the defects in this area are often accompanied by exposure of the fibula and tendons. Microsurgical tissue transfer or a pedicled flap is needed to cover those exposures for even a relatively small defect due to the insufficiency of the local cutaneous and muscle flap in this area. Koshima et al. and Wei et al. began to propose the concept of localized perforator flaps, which were initially applied to free perforator flaps. The main benefits of such localized perforator flaps are described below.

1. It preserves vital blood vessels and the underlying muscles and fascia.
2. Complications in the donor area are rare and can be direct or partial sutures.
3. Not technically demanding, although we need to find the vessel but not the vessel junction.
4. Shorter surgery time.

There are many choices of perforator flaps for lateral ankle soft tissue defects, including lateral upper ankle flap, retrograde anterior tibial artery flap, retrograde gastrocnemius flap, etc. Among them, the lateral upper ankle flap is one of the flaps commonly used for reconstruction of lateral ankle tissue defects, and the research on the lateral upper peroneal artery perforator flap is limited.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical application of the peroneal artery perforator flap with or without split-thickness skin grafting for soft tissue reconstruction of the bony defect of the lateral malleolus of the ankle joints. Reconstruction using a peroneal artery perforator flap with or without split-thickness skin grafting was performed for 10 men and 5 women patients with defects in the lateral malleolus. The mean age was 53.7 years with the age range between 22 and 89 years, and the mean size of the flaps was 40 cm^2. The soft tissue defects were caused by a diabetic foot (6 patients), infected bursitis (1 patient), chronic osteomyelitis (2 patients), and trauma (6 patients). Three of six diabetes mellitus patients also had peripheral arterial occlusive disease. The flaps were elevated in the form of a perforator flap, and split-thickness skin grafting was performed over the flaps and adjoining raw areas. The pedicled supramalleolar perforator flap is classified into two categories: (A) propeller and (B) rotation flaps. The mean follow-up duration was 30 months postsurgical.

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged 20 years old or above (including 20 years old), regardless of gender.
* Patients with lateral ankle tissue defects

Exclusion Criteria:

* The subject is aged under 20 years old.
* Patients with tissue metabolic disorders, immune dysfunction, and drug abuse.
* Patients with severe primary diseases or mental illness such as those involving the hematopoietic system, endocrine system, etc.
* Pregnant and lactating women.
* Patient who is unwilling or unable to cooperate with the trial process or follow medical advice.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 10 men and 5 women aged above 20 years old. The defects are caused by diabetes mellitus (6 subjects; 3 of them also have a peripheral arterial occlusive disease), infected bursitis (1 subject), chronic osteomyelitis (2 subjects), and trauma (6 subjects). The subjects have various comorbidity, i.e. no comorbidity (N), diabetes mellitus (DM), hypertensive cardiovascular disease (HCVD), hypertension (HTN), and peripheral arterial occlusive disease (PAOD). The defect size varies from 4 cm^2 to 25 cm^2, while the flap size varies from 9 cm^2 to 80 cm^2. The defects are located at the right or left (R or L) of the lateral malleolus of the ankle and/not at the pretibial area, or at the dorsal foot below the lateral malleolus.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Perforator flap type | 3-60 months
  The type of the flap is categorized into propeller and rotation flap. It is determined according to the distance between the perforator and the tip of the lateral malleolus. A distance of less than 2 cm used rotation-type perforator flap, while for a distance of greater than 2 cm would use propeller-type.
Flap size | 3-60 months
  The flap size is measured in the unit of cm^2. The flap size ranged from 4 cm × 3 cm to 16 cm × 6 cm.
Distance between the perforator and the tip of the lateral malleolus | 3-60 months
  The distances of all perforators from the wound, which is the tip of the lateral malleolus in this study, were measured in the unit of cm. The distance ranged from 2 cm to 5 cm.
Complication status | 3-60 months
  The complication status expresses the complication that occurred during the wound reconstruction. The status is stated as no complication (N) and the complication happened to the patients, such as "partial flap necrosis".
Follow-up month | 3-60 months
  The follow-up month indicates the duration and the follow-up of the wound reconstruction.
Donor site type | 3-60 months
  The donor site type indicates the type of skin grafting needed to be applied for covering the donor site of the patients. The donor site type in this study is divided into split-thickness skin grafting (STSG) and primary closure. The STSG was applied to 12 patients, whereas the primary closure was conducted on 3 patients.
Result status | 3-60 months
  The success of the reconstruction processes is stated in the result status. All flaps and skin graftings survived which implies all wound reconstructions were successful.

REFERENCES:
- [Background] Hallock GG. Distal lower leg local random fasciocutaneous flaps. Plast Reconstr Surg. 1990 Aug;86(2):304-11. doi: 10.1097/00006534-199008000-00018. PMID 2367579
- [Background] Koshima I, Itoh S, Nanba Y, Tsutsui T, Takahashi Y. Medial and lateral malleolar perforator flaps for repair of defects around the ankle. Ann Plast Surg. 2003 Dec;51(6):579-83. doi: 10.1097/01.sap.0000095654.07024.65. PMID 14646653
- [Background] Wei FC, Seah CS, Tsai YC, Liu SJ, Tsai MS. Fibula osteoseptocutaneous flap for reconstruction of composite mandibular defects. Plast Reconstr Surg. 1994 Feb;93(2):294-304; discussion 305-6. PMID 8310021